CLINICAL TRIAL: NCT05404451
Title: Comparison of Mulligan Mobilization Technique and Mckenzie Exercises Among Patient With Sacroilliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/515
Record Dates: First submitted 2022-05-10; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Sacroiliac Joint Somatic Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization (Experimental): Using the Technique of Mulligan Mobilization
  Interventions: Diagnostic Test: Mulligan Mobilization
- Mckenzie Exercises (Experimental): Using Mckenzie Exercises
  Interventions: Diagnostic Test: Mckenzie Exercises

INTERVENTIONS:
Diagnostic Test: Mulligan Mobilization — Using the Technique of Mulligan Mobilization
  Arms: Mulligan Mobilization
Diagnostic Test: Mckenzie Exercises — Using Mckenzie Exercises
  Arms: Mckenzie Exercises

SUMMARY:
Comparison of Mulligan Mobilization Technique and Mckenzie Exercises Among Patient with Sacroilliac Joint Dysfunction

DETAILED DESCRIPTION:
To determine comparison of mulligan mobilization technique and McKenzie exercises in patient with sacroiliac joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65.(29)
* Both male and female and Pain in low back. (17)
* Pain in sacroiliac joint (PSIS) with or without radiating to buttocks.(30)
* With acute/subacute pain within 4-12 weeks of onset and at least three of four clinical tests positive.(14)

Exclusion Criteria:

* Midline pain in back, Lumber stenosis, Lumber radiculopathy, Spondylolisthesis, Disc related pain, Pregnant females with SIJD(29),Any lower limb pathology or hip fracture, Rheumatoid arthritis(17)
* History of any orthopedic surgery, and conditions such as ankylosing spondylitis.(14)
* Spinal leminectomy
* Arthodesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Mulligan Mobilization Technique | 6 Month
  29 Participents with Mobilization applied by a therapist and an active physiological movement to end range applied by the patient. Mulligan mobilization with 10 repetitions; 3 sets. Oswestry disability questionnaire with visual analog scale (0 for minimum and 10 for Maximum pain)

SECONDARY OUTCOMES:
Mckenzie Exercises | 6 Months
  29 Participents with intervention technique Lie down on your stomach. Prop yourself up on your forearms with your shoulders above your elbows, Hold for 2 to 3 minutes, Lower your upper body. Repeat up to eight times a day. Modified Oswestry disability questionnaire with visual analog scale(0 for minimum and 10 for Maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Social Security hospital Manga road Raiwind.,Chaudary Muhammad Akram research and teaching hospital., Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No